CLINICAL TRIAL: NCT00559832
Title: Prevention of Acute Mountain Sickness by Sleeping at Simulated Altitude (Normobaric Hypoxia)
Brief Title: Prevention of Acute Mountain Sickness by Intermittent Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 039/2006
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-11

CONDITIONS: Acute Mountain Sickness
Keywords: acute mountain sickness; intermittent hypoxia; acclimatization
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normoxia (No Intervention): Sleeping in normoxia for 14 nights prior to one night at 4500 m
- Hypoxia (Experimental): Sleeping in normobaric hypoxia for 14 nights at altitudes from 2500 - 3300 m prior to one night at 4500 m
  Interventions: Other: Hypoxic Exposure

INTERVENTIONS:
Other: Hypoxic Exposure — Sleeping in normobaric hypoxia for 14 nights at altitudes from 2500 - 3300 m prior to one night at 4500 m
  Arms: Hypoxia

SUMMARY:
Acclimatization by mountaineering prior to high altitude sojourns have shown to be effective in prevention of acute mountain sickness (AMS).

The aim of this study is to investigate whether intermittent exposure to normobaric hypoxia during sleep is also effective to prevent AMS.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* Altitude exposure above 2000 m 8 weeks prior or during the study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2006-03; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
incidence of acute mountain sickness | during one night at 4500 m

SECONDARY OUTCOMES:
Sleep quality | during one night at altitude
ventilatory acclimatization | during one night at altitude

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Dehnert, MD, Principal Investigator — University Hospital Heidelberg
Locations (1):
- Sports Medicine, University Hospital, Heidelberg, Germany